CLINICAL TRIAL: NCT04802707
Title: A Phase II, Monocenter, Single Arm Study To Assess The Safety and Efficacy Of Combination Deoxycytidine and Deoxythymidine For Mitochondrial Depletion Disorders
Brief Title: Deoxynucleosides Pyrimidines as Treatment for Mitochondrial Depletion Syndrome
Acronym: dC-dT-MDS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kenneth Myers, MD (Other)
Responsible Party: Sponsor-Investigator, Kenneth Myers, MD, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-7654 dC-dT-MDS
Record Dates: First submitted 2021-03-10; First posted 2021-03-17 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Mitochondrial Diseases; Mitochondrial Encephalomyopathy; Mitochondrial Encephalopathy; Mitochondrial DNA Depletion; Mitochondrial Metabolism Disorders
Keywords: Deoxycytidine; Deoxythymidine; Deoxynucleoside; Pyrimidine; Mitochondria; mtDNA; Depletion
MeSH Terms: conditions — Mitochondrial Diseases; Mitochondrial Encephalomyopathies; Mitochondrial encephalopathy | interventions — Deoxycytidine; Thymidine

STUDY DESIGN:
Intervention Model Description: Phase II, One Site, Open label study in the pediatric and adult population
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dC/dT100-400 Arm (Experimental): Children & Adult (0-60 Y), who takes the investigational product deoxynucleosides pyrimidine (mix of deoxycytidine and deoxythymidine), following the protocol.
  Interventions: Combination Product: deoxycytidine and deoxythymidine

INTERVENTIONS:
Combination Product: deoxycytidine and deoxythymidine — The Investigational Product (IP) dC/dT100-400 will be administered orally every day (QD) and the dose is divided over trid or bid for the daily dose of 100 mg/kg from Day 1-7, 200 mg/kg from Day 8-14, 300 mg/kg from Day 15- 21 and 400 mg/kg from Day 22 to 1825. Doses was chosen according to the safety and efficacy doses used in the literature.

SUMMARY:
Mitochondrial DNA (mtDNA) depletion syndromes (MDS) are a genetically and clinically heterogeneous group of autosomal recessive disorders that are characterized by a severe reduction in mtDNA content leading to impaired energy production in affected tissues and organs. MDS are due to defects in mtDNA maintenance caused by mutations in nuclear genes that function in either mitochondrial nucleotide synthesis. MDS are phenotypically heterogeneous and usually classified as myopathic, encephalomyopathic, hepatocerebral or neurogastrointestinal.

No efficacious therapy is available for any of these disorders. Affected individuals should have a comprehensive evaluation to assess the degree of involvement of different systems. Treatment is directed mainly toward providing symptomatic management. No treatment for MDS.

Clinical trials studies and in vitro/in vivo research studies showed that the enhancement of the salvage pathway by increasing the availability of deoxyribonucleosides needed for each specific genetic defect prevents mtDNA depletion.

Early recognition and immediate therapy to restore mitochondrial function could potentially improve clinical course.

Confirming the benefit of deoxynucleosides as a safe and potentially efficacious therapy, will lead to the availability of the first specific and effective treatment for Mitochondria Depletion Disorders.

In this phase II Trial a mix of Deoxynucleosides Pyrimidine (Deoxycytidine dC and Deoxythymidine dT) will be used as early treatment of MDS.

The dose used has been already used in other clinical trials, and appears to effective and well-tolerated. The subjects included are children (0-18Y), with positive MDS diagnosis and express mutations in one of the following genes: POLG, POLG2, C10orf2, RRM2B, MPV17, SUCLA2, SUCLG1, FBXL4, DTYMK. Subjects with MDS expressing neurological phenotypes dysfunction.

DETAILED DESCRIPTION:
This Trial is designed as Phase II, Monocenter, Open label study in the pediatric population.

The aim is to evaluate the safety, tolerability and efficacy of Deoxycytidine and Deoxythymidine in treatment of children with Mitochondrial Depletion Disorders.

Primary Objectives The primary objective of this study is to evaluate the efficacy of dC/dT100-400 in subjects with mitochondria depletion disorders.

Secondary Objectives The secondary objectives of this study are to evaluate tolerability and safety of dC/dT100-400 in subjects with mitochondria depletion disorders.

Efficacy of dC/dT100-400 :

First Outcomes:

1. Improved clinical status observed during the genetic follow-up and the Newcastle Paediatric Mitochondrial Disease Scale (NPMDS) or Adult Newcastle Mitochondrial Disease Scale (ANMDS), which are validated measures used by geneticists to allow evaluation of the progression of mitochondrial disease in patients 0-60 y.
2. Evaluation of growth differentiation factor 15 (GDF15; a marker of severity of mitochondria dysfunction).

Secondary Outcomes:

1. Safety and tolerability will be tested by recording adverse effects (AE): AE will be monitored and collected throughout the study.

   * Diarrhea: Reported diarrhea frequency during the treatment, will permit to define the tolerability of dC/dT100-400.
   * AE leading to study drug discontinuation, treatment-emergent adverse events (TEAEs), SAEs (Severe Adverse Effect) will be reported from the first day the subjects start taking medication until the last dose taken.
2. Neurological improvement by electroencephalography (EEG), seizure diary, development and quality of life questionnaires (PED and adults), clinical status observed during the neurological follow-up.
3. Bloodwork for different assessments:

   Complete blood and platelet counts (CBC) will be performed to monitor any potential toxicity, liver function (aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), bilirubin and albumin.), kidney function (creatinine, urea, electrolytes). Assess for myopathy with serum creatine kinase (CK).
4. mtDNA quantification.
5. Evaluation of mitochondrial function with capillary/venous blood gas, serum lactate, plasma amino acids, acylcarnitine profile, urine amino acids, urine purines and pyrimidines acids.

ELIGIBILITY:
Inclusion Criteria:

* Children & Adults (0 -60 Y)
* Written informed consent obtained,
* Clinical Diagnosis of a Mitochondrial Depletion Disorder.
* Pathogenic variant(s) Homozygote and Heterozygote in one of the following genes: POLG, POLG2, C10orf2, RRM2B, MPV17, SUCLA2, SUCLG1, FBXL4, DTYMK
* Females of childbearing age:

Negative urinary pregnancy test at screening Agree to use effective contraception for the duration of the study

Exclusion Criteria:

* Inability of a parent or legal guardian to give informed consent for any reason
* Chronic severe diarrhea

Ages: 1 Month to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Responder versus Non-Responder Status with investigational product | 260 weeks
  There is no estimation of sample size, the number will depend on subjects enrolled. We assume we can include about 50 to 100 subjects with mitochondrial depletion disorder. This study is designed as Phase II trial case series, the data will be presented graphically The IP of study will be considered positive if more than 2 responders are observed in 5 subjects. This design yields a marginal one-sided type I error rate (α) of 5% and power of 80%. For more than one participant engages in a study, the spaghetti plot showing all of their data in the same figure will be used as tool for visualization. Visual analysis of graphed data has been the traditional method for evaluating treatment effects in series cases research.

SECONDARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities, adverse events (AEs), serious adverse events (SAEs) | 260 weeks
  "Responder" defined as having ≥ 2 of (1) electroencephalography EEG improvement, (2) decreased seizure frequency, (3) cognitive improvement, (4) caregiver impression of improvement, (5) clinical improvement, (6) Safety profile will be assessed through number of participants experiencing adverse events (AEs), serious adverse events (SAEs), laboratory evaluations, vital signs, and physical examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Alexis MD Myers, MD PhD FRCPC, Principal Investigator — RI-MUHC, Children Hospital of Montreal (MUHC), McGill University
Locations (1):
- Research InstituMcGill University Health Centre - Children Hospital of Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
REDCap software will be used as IPD. The data's will be shared anonymous, subject will bes identified by an Identifiant (ID).
  REDCap is managed by quality data's teams of research institute of McGill University Health Center (RI-MUHC).
  For clinical study reports since the study is planned at the Children Hospital of Montreal, Clinical Study Report (CSR) access will be done through open architecture clinical information system (Oacis) tool of hospital Study Protocol And Informed Consent Form (ICF) will be shared by Email or on core network of RIMUHC
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 104 weeks
Access Criteria: Research Staff, Principal Investigator (PI), Co-Investigator, regulation authority and clinical research associate (CRA) for monitoring are authorized to access to the data's for CRA (anonymous data's)

REFERENCES:
- [Background] Osellame LD, Blacker TS, Duchen MR. Cellular and molecular mechanisms of mitochondrial function. Best Pract Res Clin Endocrinol Metab. 2012 Dec;26(6):711-23. doi: 10.1016/j.beem.2012.05.003. Epub 2012 Jun 23. PMID 23168274
- [Background] Miller FJ, Rosenfeldt FL, Zhang C, Linnane AW, Nagley P. Precise determination of mitochondrial DNA copy number in human skeletal and cardiac muscle by a PCR-based assay: lack of change of copy number with age. Nucleic Acids Res. 2003 Jun 1;31(11):e61. doi: 10.1093/nar/gng060. PMID 12771225
- [Background] DiMauro S, Schon EA. Mitochondrial respiratory-chain diseases. N Engl J Med. 2003 Jun 26;348(26):2656-68. doi: 10.1056/NEJMra022567. No abstract available. PMID 12826641
- [Background] Huang CC, Hsu CH. [Mitochondrial disease and mitochondrial DNA depletion syndromes]. Acta Neurol Taiwan. 2009 Dec;18(4):287-95. Chinese. PMID 20329599
- [Background] Rusecka J, Kaliszewska M, Bartnik E, Tonska K. Nuclear genes involved in mitochondrial diseases caused by instability of mitochondrial DNA. J Appl Genet. 2018 Feb;59(1):43-57. doi: 10.1007/s13353-017-0424-3. Epub 2018 Jan 17. PMID 29344903
- [Background] Viscomi C, Zeviani M. MtDNA-maintenance defects: syndromes and genes. J Inherit Metab Dis. 2017 Jul;40(4):587-599. doi: 10.1007/s10545-017-0027-5. Epub 2017 Mar 21. PMID 28324239
- [Background] Blazquez-Bermejo C, Carreno-Gago L, Molina-Granada D, Aguirre J, Ramon J, Torres-Torronteras J, Cabrera-Perez R, Martin MA, Dominguez-Gonzalez C, de la Cruz X, Lombes A, Garcia-Arumi E, Marti R, Camara Y. Increased dNTP pools rescue mtDNA depletion in human POLG-deficient fibroblasts. FASEB J. 2019 Jun;33(6):7168-7179. doi: 10.1096/fj.201801591R. Epub 2019 Mar 8. PMID 30848931
- [Background] El-Hattab AW, Scaglia F. Mitochondrial DNA depletion syndromes: review and updates of genetic basis, manifestations, and therapeutic options. Neurotherapeutics. 2013 Apr;10(2):186-98. doi: 10.1007/s13311-013-0177-6. PMID 23385875
- [Background] Nogueira C, Almeida LS, Nesti C, Pezzini I, Videira A, Vilarinho L, Santorelli FM. Syndromes associated with mitochondrial DNA depletion. Ital J Pediatr. 2014 Apr 3;40:34. doi: 10.1186/1824-7288-40-34. PMID 24708634
- [Background] Basel D. Mitochondrial DNA Depletion Syndromes. Clin Perinatol. 2020 Mar;47(1):123-141. doi: 10.1016/j.clp.2019.10.008. Epub 2019 Oct 31. PMID 32000920
- [Background] Rahman S, Poulton J. Diagnosis of mitochondrial DNA depletion syndromes. Arch Dis Child. 2009 Jan;94(1):3-5. doi: 10.1136/adc.2008.147983. No abstract available. PMID 19103785
- [Background] Spinazzola A, Invernizzi F, Carrara F, Lamantea E, Donati A, Dirocco M, Giordano I, Meznaric-Petrusa M, Baruffini E, Ferrero I, Zeviani M. Clinical and molecular features of mitochondrial DNA depletion syndromes. J Inherit Metab Dis. 2009 Apr;32(2):143-58. doi: 10.1007/s10545-008-1038-z. Epub 2008 Dec 27. PMID 19125351
- [Background] Suomalainen A, Isohanni P. Mitochondrial DNA depletion syndromes--many genes, common mechanisms. Neuromuscul Disord. 2010 Jul;20(7):429-37. doi: 10.1016/j.nmd.2010.03.017. Epub 2010 May 4. PMID 20444604
- [Background] Copeland WC. Defects in mitochondrial DNA replication and human disease. Crit Rev Biochem Mol Biol. 2012 Jan-Feb;47(1):64-74. doi: 10.3109/10409238.2011.632763. PMID 22176657
- [Background] Khan NA, Govindaraj P, Meena AK, Thangaraj K. Mitochondrial disorders: challenges in diagnosis & treatment. Indian J Med Res. 2015 Jan;141(1):13-26. doi: 10.4103/0971-5916.154489. PMID 25857492
- [Background] Hikmat O, Eichele T, Tzoulis C, Bindoff LA. Understanding the Epilepsy in POLG Related Disease. Int J Mol Sci. 2017 Aug 24;18(9):1845. doi: 10.3390/ijms18091845. PMID 28837072
- [Background] El-Hattab AW, Craigen WJ, Scaglia F. Mitochondrial DNA maintenance defects. Biochim Biophys Acta Mol Basis Dis. 2017 Jun;1863(6):1539-1555. doi: 10.1016/j.bbadis.2017.02.017. Epub 2017 Feb 16. PMID 28215579
- [Background] El-Hattab AW, Craigen WJ, Wong LJC, Scaglia F. Mitochondrial DNA Maintenance Defects Overview. 2018 Mar 8. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK487393/ PMID 29517884
- [Background] Copeland WC. Defects of mitochondrial DNA replication. J Child Neurol. 2014 Sep;29(9):1216-24. doi: 10.1177/0883073814537380. Epub 2014 Jun 30. PMID 24985751
- [Background] Spinazzola A, Zeviani M. Disorders from perturbations of nuclear-mitochondrial intergenomic cross-talk. J Intern Med. 2009 Feb;265(2):174-92. doi: 10.1111/j.1365-2796.2008.02059.x. PMID 19192035
- [Background] Cohen, B.H., P.F. Chinnery, and W.C. Copeland, POLG-Related Disorders, in GeneReviews((R)), M.P. Adam, et al., Editors. 1993: Seattle (WA).
- [Background] Milone M, Benarroch EE, Wong LJ. POLG-related disorders: defects of the nuclear and mitochondrial genome interaction. Neurology. 2011 Nov 15;77(20):1847-52. doi: 10.1212/WNL.0b013e318238863a. No abstract available. PMID 22084276
- [Background] Rahman S, Copeland WC. POLG-related disorders and their neurological manifestations. Nat Rev Neurol. 2019 Jan;15(1):40-52. doi: 10.1038/s41582-018-0101-0. PMID 30451971
- [Background] Anagnostou ME, Ng YS, Taylor RW, McFarland R. Epilepsy due to mutations in the mitochondrial polymerase gamma (POLG) gene: A clinical and molecular genetic review. Epilepsia. 2016 Oct;57(10):1531-1545. doi: 10.1111/epi.13508. Epub 2016 Aug 24. PMID 27554452
- [Background] Engelsen BA, Tzoulis C, Karlsen B, Lillebo A, Laegreid LM, Aasly J, Zeviani M, Bindoff LA. POLG1 mutations cause a syndromic epilepsy with occipital lobe predilection. Brain. 2008 Mar;131(Pt 3):818-28. doi: 10.1093/brain/awn007. Epub 2008 Jan 30. PMID 18238797
- [Background] Horvath R, Hudson G, Ferrari G, Futterer N, Ahola S, Lamantea E, Prokisch H, Lochmuller H, McFarland R, Ramesh V, Klopstock T, Freisinger P, Salvi F, Mayr JA, Santer R, Tesarova M, Zeman J, Udd B, Taylor RW, Turnbull D, Hanna M, Fialho D, Suomalainen A, Zeviani M, Chinnery PF. Phenotypic spectrum associated with mutations of the mitochondrial polymerase gamma gene. Brain. 2006 Jul;129(Pt 7):1674-84. doi: 10.1093/brain/awl088. Epub 2006 Apr 18. PMID 16621917
- [Background] Hikmat O, Tzoulis C, Chong WK, Chentouf L, Klingenberg C, Fratter C, Carr LJ, Prabhakar P, Kumaraguru N, Gissen P, Cross JH, Jacques TS, Taanman JW, Bindoff LA, Rahman S. Correction: The clinical spectrum and natural history of early-onset diseases due to DNA polymerase gamma mutations. Genet Med. 2019 Apr;21(4):1027. doi: 10.1038/s41436-018-0098-1. PMID 30228318
- [Background] Lim A, Thomas RH. The mitochondrial epilepsies. Eur J Paediatr Neurol. 2020 Jan;24:47-52. doi: 10.1016/j.ejpn.2019.12.021. Epub 2020 Jan 7. PMID 31973983
- [Background] Ashley N, Adams S, Slama A, Zeviani M, Suomalainen A, Andreu AL, Naviaux RK, Poulton J. Defects in maintenance of mitochondrial DNA are associated with intramitochondrial nucleotide imbalances. Hum Mol Genet. 2007 Jun 15;16(12):1400-11. doi: 10.1093/hmg/ddm090. Epub 2007 May 3. PMID 17483096
- [Background] Gandhi VV, Samuels DC. A review comparing deoxyribonucleoside triphosphate (dNTP) concentrations in the mitochondrial and cytoplasmic compartments of normal and transformed cells. Nucleosides Nucleotides Nucleic Acids. 2011 May;30(5):317-39. doi: 10.1080/15257770.2011.586955. PMID 21774628
- [Background] Gonzalez-Vioque E, Torres-Torronteras J, Andreu AL, Marti R. Limited dCTP availability accounts for mitochondrial DNA depletion in mitochondrial neurogastrointestinal encephalomyopathy (MNGIE). PLoS Genet. 2011 Mar;7(3):e1002035. doi: 10.1371/journal.pgen.1002035. Epub 2011 Mar 31. PMID 21483760
- [Background] Absalon MJ, Harding CO, Fain DR, Li L, Mack KJ. Leigh syndrome in an infant resulting from mitochondrial DNA depletion. Pediatr Neurol. 2001 Jan;24(1):60-3. doi: 10.1016/s0887-8994(00)00226-5. PMID 11182283
- [Background] Keshavan N, Abdenur J, Anderson G, Assouline Z, Barcia G, Bouhikbar L, Chakrapani A, Cleary M, Cohen MC, Feillet F, Fratter C, Hauser N, Jacques T, Lam A, McCullagh H, Phadke R, Rotig A, Sharrard M, Simon M, Smith C, Sommerville EW, Taylor RW, Yue WW, Rahman S. The natural history of infantile mitochondrial DNA depletion syndrome due to RRM2B deficiency. Genet Med. 2020 Jan;22(1):199-209. doi: 10.1038/s41436-019-0613-z. Epub 2019 Aug 29. PMID 31462754
- [Background] Shaibani A, Shchelochkov OA, Zhang S, Katsonis P, Lichtarge O, Wong LJ, Shinawi M. Mitochondrial neurogastrointestinal encephalopathy due to mutations in RRM2B. Arch Neurol. 2009 Aug;66(8):1028-32. doi: 10.1001/archneurol.2009.139. PMID 19667227
- [Background] Bourdon A, Minai L, Serre V, Jais JP, Sarzi E, Aubert S, Chretien D, de Lonlay P, Paquis-Flucklinger V, Arakawa H, Nakamura Y, Munnich A, Rotig A. Mutation of RRM2B, encoding p53-controlled ribonucleotide reductase (p53R2), causes severe mitochondrial DNA depletion. Nat Genet. 2007 Jun;39(6):776-80. doi: 10.1038/ng2040. Epub 2007 May 7. PMID 17486094
- [Background] Kollberg G, Darin N, Benan K, Moslemi AR, Lindal S, Tulinius M, Oldfors A, Holme E. A novel homozygous RRM2B missense mutation in association with severe mtDNA depletion. Neuromuscul Disord. 2009 Feb;19(2):147-50. doi: 10.1016/j.nmd.2008.11.014. Epub 2009 Jan 12. PMID 19138848
- [Background] El-Hattab AW, Wang J, Dai H, Almannai M, Scaglia F, Craigen WJ, Wong LJC. MPV17-Related Mitochondrial DNA Maintenance Defect. 2012 May 17 [updated 2018 May 17]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK92947/ PMID 22593919
- [Background] El-Hattab AW, Wang J, Dai H, Almannai M, Staufner C, Alfadhel M, Gambello MJ, Prasun P, Raza S, Lyons HJ, Afqi M, Saleh MAM, Faqeih EA, Alzaidan HI, Alshenqiti A, Flore LA, Hertecant J, Sacharow S, Barbouth DS, Murayama K, Shah AA, Lin HC, Wong LC. MPV17-related mitochondrial DNA maintenance defect: New cases and review of clinical, biochemical, and molecular aspects. Hum Mutat. 2018 Apr;39(4):461-470. doi: 10.1002/humu.23387. Epub 2018 Jan 13. PMID 29282788
- [Background] El-Hattab AW, Scaglia F. SUCLA2-Related Mitochondrial DNA Depletion Syndrome, Encephalomyopathic Form with Methylmalonic Aciduria. 2009 May 26 [updated 2023 Sep 28]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK6803/ PMID 20301762
- [Background] El-Hattab AW, Scaglia F. SUCLG1-Related Mitochondrial DNA Depletion Syndrome, Encephalomyopathic Form with Methylmalonic Aciduria. 2017 Mar 30. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK425223/ PMID 28358460
- [Background] Almannai M, Dai H, El-Hattab AW, Wong LJC. FBXL4-Related Encephalomyopathic Mitochondrial DNA Depletion Syndrome. 2017 Apr 6. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK425540/ PMID 28383868
- [Background] Saada A. Deoxyribonucleotides and disorders of mitochondrial DNA integrity. DNA Cell Biol. 2004 Dec;23(12):797-806. doi: 10.1089/dna.2004.23.797. PMID 15684706
- [Background] Wang L. Mitochondrial purine and pyrimidine metabolism and beyond. Nucleosides Nucleotides Nucleic Acids. 2016 Dec;35(10-12):578-594. doi: 10.1080/15257770.2015.1125001. PMID 27906631
- [Background] Akanuma J. [Mitochondrial DNA depletion syndrome]. Nihon Rinsho. 2002 Apr;60 Suppl 4:398-401. No abstract available. Japanese. PMID 12013896
- [Background] Zipursky A. The genetics of childhood disease and development. Pediatr Res. 2003 Jan;53(1):3. doi: 10.1203/00006450-200301000-00003. No abstract available. PMID 12508073
- [Background] Filosto M, Scarpelli M, Tonin P, Lucchini G, Pavan F, Santus F, Parini R, Donati MA, Cotelli MS, Vielmi V, Todeschini A, Canonico F, Tomelleri G, Padovani A, Rovelli A. Course and management of allogeneic stem cell transplantation in patients with mitochondrial neurogastrointestinal encephalomyopathy. J Neurol. 2012 Dec;259(12):2699-706. doi: 10.1007/s00415-012-6572-9. Epub 2012 Jun 19. PMID 22711161
- [Background] Hirano M, Marti R, Casali C, Tadesse S, Uldrick T, Fine B, Escolar DM, Valentino ML, Nishino I, Hesdorffer C, Schwartz J, Hawks RG, Martone DL, Cairo MS, DiMauro S, Stanzani M, Garvin JH Jr, Savage DG. Allogeneic stem cell transplantation corrects biochemical derangements in MNGIE. Neurology. 2006 Oct 24;67(8):1458-60. doi: 10.1212/01.wnl.0000240853.97716.24. Epub 2006 Sep 13. PMID 16971696
- [Background] Yavuz H, Ozel A, Christensen M, Christensen E, Schwartz M, Elmaci M, Vissing J. Treatment of mitochondrial neurogastrointestinal encephalomyopathy with dialysis. Arch Neurol. 2007 Mar;64(3):435-8. doi: 10.1001/archneur.64.3.435. PMID 17353390
- [Background] Hasselmann O, Blau N, Ramaekers VT, Quadros EV, Sequeira JM, Weissert M. Cerebral folate deficiency and CNS inflammatory markers in Alpers disease. Mol Genet Metab. 2010 Jan;99(1):58-61. doi: 10.1016/j.ymgme.2009.08.005. PMID 19766516
- [Background] Rodriguez MC, MacDonald JR, Mahoney DJ, Parise G, Beal MF, Tarnopolsky MA. Beneficial effects of creatine, CoQ10, and lipoic acid in mitochondrial disorders. Muscle Nerve. 2007 Feb;35(2):235-42. doi: 10.1002/mus.20688. PMID 17080429
- [Background] Saito K, Kimura N, Oda N, Shimomura H, Kumada T, Miyajima T, Murayama K, Tanaka M, Fujii T. Pyruvate therapy for mitochondrial DNA depletion syndrome. Biochim Biophys Acta. 2012 May;1820(5):632-6. doi: 10.1016/j.bbagen.2011.08.006. Epub 2011 Aug 11. PMID 21855607
- [Background] Wong LJ, Naviaux RK, Brunetti-Pierri N, Zhang Q, Schmitt ES, Truong C, Milone M, Cohen BH, Wical B, Ganesh J, Basinger AA, Burton BK, Swoboda K, Gilbert DL, Vanderver A, Saneto RP, Maranda B, Arnold G, Abdenur JE, Waters PJ, Copeland WC. Molecular and clinical genetics of mitochondrial diseases due to POLG mutations. Hum Mutat. 2008 Sep;29(9):E150-72. doi: 10.1002/humu.20824. PMID 18546365
- [Background] Lara MC, Valentino ML, Torres-Torronteras J, Hirano M, Marti R. Mitochondrial neurogastrointestinal encephalomyopathy (MNGIE): biochemical features and therapeutic approaches. Biosci Rep. 2007 Jun;27(1-3):151-63. doi: 10.1007/s10540-007-9043-2. PMID 17549623
- [Background] Lara MC, Weiss B, Illa I, Madoz P, Massuet L, Andreu AL, Valentino ML, Anikster Y, Hirano M, Marti R. Infusion of platelets transiently reduces nucleoside overload in MNGIE. Neurology. 2006 Oct 24;67(8):1461-3. doi: 10.1212/01.wnl.0000239824.95411.52. Epub 2006 Sep 13. PMID 16971699
- [Background] Camara Y, Gonzalez-Vioque E, Scarpelli M, Torres-Torronteras J, Marti R. Feeding the deoxyribonucleoside salvage pathway to rescue mitochondrial DNA. Drug Discov Today. 2013 Oct;18(19-20):950-7. doi: 10.1016/j.drudis.2013.06.009. Epub 2013 Jun 28. PMID 23817075
- [Background] Uusimaa J, Evans J, Smith C, Butterworth A, Craig K, Ashley N, Liao C, Carver J, Diot A, Macleod L, Hargreaves I, Al-Hussaini A, Faqeih E, Asery A, Al Balwi M, Eyaid W, Al-Sunaid A, Kelly D, van Mourik I, Ball S, Jarvis J, Mulay A, Hadzic N, Samyn M, Baker A, Rahman S, Stewart H, Morris AA, Seller A, Fratter C, Taylor RW, Poulton J. Clinical, biochemical, cellular and molecular characterization of mitochondrial DNA depletion syndrome due to novel mutations in the MPV17 gene. Eur J Hum Genet. 2014 Feb;22(2):184-91. doi: 10.1038/ejhg.2013.112. Epub 2013 May 29. PMID 23714749
- [Background] Dalla Rosa I, Camara Y, Durigon R, Moss CF, Vidoni S, Akman G, Hunt L, Johnson MA, Grocott S, Wang L, Thorburn DR, Hirano M, Poulton J, Taylor RW, Elgar G, Marti R, Voshol P, Holt IJ, Spinazzola A. MPV17 Loss Causes Deoxynucleotide Insufficiency and Slow DNA Replication in Mitochondria. PLoS Genet. 2016 Jan 13;12(1):e1005779. doi: 10.1371/journal.pgen.1005779. eCollection 2016 Jan. PMID 26760297
- [Background] Bulst S, Holinski-Feder E, Payne B, Abicht A, Krause S, Lochmuller H, Chinnery PF, Walter MC, Horvath R. In vitro supplementation with deoxynucleoside monophosphates rescues mitochondrial DNA depletion. Mol Genet Metab. 2012 Sep;107(1-2):95-103. doi: 10.1016/j.ymgme.2012.04.022. Epub 2012 May 3. PMID 22608879
- [Background] Franzolin E, Salata C, Bianchi V, Rampazzo C. The Deoxynucleoside Triphosphate Triphosphohydrolase Activity of SAMHD1 Protein Contributes to the Mitochondrial DNA Depletion Associated with Genetic Deficiency of Deoxyguanosine Kinase. J Biol Chem. 2015 Oct 23;290(43):25986-96. doi: 10.1074/jbc.M115.675082. Epub 2015 Sep 4. PMID 26342080
- [Background] Akman HO, Dorado B, Lopez LC, Garcia-Cazorla A, Vila MR, Tanabe LM, Dauer WT, Bonilla E, Tanji K, Hirano M. Thymidine kinase 2 (H126N) knockin mice show the essential role of balanced deoxynucleotide pools for mitochondrial DNA maintenance. Hum Mol Genet. 2008 Aug 15;17(16):2433-40. doi: 10.1093/hmg/ddn143. Epub 2008 May 8. PMID 18467430
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Background] Dominguez-Gonzalez C, Madruga-Garrido M, Mavillard F, Garone C, Aguirre-Rodriguez FJ, Donati MA, Kleinsteuber K, Marti I, Martin-Hernandez E, Morealejo-Aycinena JP, Munell F, Nascimento A, Kalko SG, Sardina MD, Alvarez Del Vayo C, Serrano O, Long Y, Tu Y, Levin B, Thompson JLP, Engelstad K, Uddin J, Torres-Torronteras J, Jimenez-Mallebrera C, Marti R, Paradas C, Hirano M. Deoxynucleoside Therapy for Thymidine Kinase 2-Deficient Myopathy. Ann Neurol. 2019 Aug;86(2):293-303. doi: 10.1002/ana.25506. Epub 2019 Jun 17. PMID 31125140
- [Background] Hernandez-Voth A, Sayas Catalan J, Corral Blanco M, Castano Mendez A, Martin MA, De Fuenmayor Fernandez de la Hoz C, Villena Garrido V, Dominguez-Gonzalez C. Deoxynucleoside therapy for respiratory involvement in adult patients with thymidine kinase 2-deficient myopathy. BMJ Open Respir Res. 2020 Nov;7(1):e000774. doi: 10.1136/bmjresp-2020-000774. PMID 33246973
- [Background] Purine and pyrimidine metabolism. Ciba Found Symp. 1977;(48):331-55. No abstract available. PMID 245993
- [Background] Bory C, Chantin C, Boulieu R. Abnormal purine and pyrimidine metabolism in inherited superactivity of PRPP synthetase. Adv Exp Med Biol. 1994;370:15-8. doi: 10.1007/978-1-4615-2584-4_4. No abstract available. PMID 7660879
- [Background] Castellanos M, Wilson DB, Shuler ML. A modular minimal cell model: purine and pyrimidine transport and metabolism. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6681-6. doi: 10.1073/pnas.0400962101. Epub 2004 Apr 16. PMID 15090651
- [Background] Khan I, Sarker SJ, Hackshaw A. Smaller sample sizes for phase II trials based on exact tests with actual error rates by trading-off their nominal levels of significance and power. Br J Cancer. 2012 Nov 20;107(11):1801-9. doi: 10.1038/bjc.2012.444. PMID 23169334
- [Derived] Pekeles H, Berrahmoune S, Dassi C, Cheung ACT, Gagnon T, Waters PJ, Eberhard R, Buhas D, Myers KA. Safety and efficacy of deoxycytidine/deoxythymidine combination therapy in POLG-related disorders: 6-month interim results of an open-label, single arm, phase 2 trial. EClinicalMedicine. 2024 Jul 18;74:102740. doi: 10.1016/j.eclinm.2024.102740. eCollection 2024 Aug. PMID 39091670